CLINICAL TRIAL: NCT01268319
Title: A Randomized Pilot Trial of the Use of a Distal Protection Device to Prevent Peri-procedural MI During Dilation of Coronary Stenoses Caused by Plaques With Large Lipid Cores
Brief Title: CANARY: Coronary Assessment by Near-infrared of Atherosclerotic Rupture-prone Yellow
Acronym: CANARY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Infraredx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0114
Record Dates: First submitted 2010-12-28; First posted 2010-12-30 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Coronary Atherosclerosis; Myocardial Infarction; Coronary Plaque Embolization
Keywords: Myocardial Infarction; percutaneous coronary intervention; embolization; necrotic core; vulnerable plaque; coronary plaque rupture
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Embolic Protection Devices; Angioplasty; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- (+)HR-LCP and EPD (Experimental): These subjects will meet all angiographic criteria.The target plaque will contain a LipiScan IVUS signal that meets the Higher Risk Lipid Core Plaque (HR-LCP) definition contained in the protocol. 27 Subjects who meet this criteria will be randomized to standard pre-dilation and stent implantation with an embolic protection device (EPD)in place prior to any angioplasty.
  Interventions: Device: Embolic Protection Device (EPD); Device: Intracoronary Spectroscopy and Ultrasonic Evaluation; Device: Angioplasty and Stent Implant
- (+)HR-LCP and No EPD (standard of care) (Placebo Comparator): These subjects will meet all angiographic criteria.The target plaque will contain a LipiScan IVUS signal that meets the Higher Risk Lipid Core Plaque (HR-LCP) definition contained in the protocol. 27 Subjects who meet this criteria will be randomized to standard pre-dilation and stent implantation without an embolic protection device (EPD)in place prior to any angioplasty.
  Interventions: Device: Intracoronary Spectroscopy and Ultrasonic Evaluation; Device: Angioplasty and Stent Implant
- (-)HR-LCP and No EPD (standard of care) (Placebo Comparator): These subjects will meet all angiographic criteria.The target plaque will NOT contain a LipiScan IVUS signal that meets the Higher Risk Lipid Core Plaque (HR-LCP) definition contained in the protocol. 54 Subjects who meet this criteria will be assigned (not randomized) to standard pre-dilation and stent implantation without an embolic protection device (EPD)in place prior to any angioplasty.
  Interventions: Device: Intracoronary Spectroscopy and Ultrasonic Evaluation; Device: Angioplasty and Stent Implant

INTERVENTIONS:
Device: Embolic Protection Device (EPD) — The embolic protection device consists of a protection wire, a delivery sheath, a retrieval sheath and various accessories (wire torque device, introducer, dilator tool). The wire of the EPD is used as a standard 0.014" steerable guide wire. The filter is designed for embolic debris capture while maintaining continuous blood flow. At the completion of the procedure, the filter and its contents are removed using the retrieval sheath and then removed from the patient.
  Other Names: Filterwire
  Arms: (+)HR-LCP and EPD
Device: Intracoronary Spectroscopy and Ultrasonic Evaluation — This intervention requires a near infrared imaging catheter equipped with an intravascular ultrasonic transducer be used to evaluate the coronary artery wall prior to treatment and after treatment. This system detects the lipid containing plaques that may be the source of embolic debris released during standard angioplasty and stent placement.
  Other Names: LipiScan IVUS Coronary Imaging System; LipiScan IVUS; LipiScan; Chemogram
Device: Angioplasty and Stent Implant — The target plaque will be treated with a pre-dilation with a standard angioplasty balloon sized to within 0.5mm of the diameter of the reference vessel diameter. The physician will then implant a coronary artery stent that is appropriately sized for the reference vessel diameter.

SUMMARY:
The CANARY (Coronary Assessment by Near-infrared of Atherosclerotic Rupture-prone Yellow) Study is a pivotal trial to evaluate criteria for defining a Lipid Core Plaque (LCP) that is at high risk of rupturing during standard of care therapy and causing intra-procedural complications. If plaques that require treatment are at higher than normal risk of causing intra-procedural complications, some life threatening, the treating physician is better informed and may opt to take precautionary measures to mitigate the risk or result of a complication. The CANARY Study is also designed to evaluate the feasibility of using a distal embolization protection device (EPD) as a means to prevent heart attacks triggered by the embolization of plaque during standard care therapy. It is thought that the EPD will prevent plaque from going downstream during treatment and obstructing other heart vessels. These obstructions could cause heart attacks by preventing blood from reaching heart muscle tissue.

ELIGIBILITY:
Inclusion Criteria

* Subject is at least 18 years of age
* Subject is scheduled for an elective coronary catheterization
* Subject is willing and able to provide informed written consent prior to the index catheterization
* LipiScan IVUS CIS use is not contra-indicated
* At least one submitted Chemogram is obtained entirely within a native coronary artery
* Patient has been diagnosed with: stable angina (CCS I or CCS II);a positive functional test for ischemia (within the preceding 30 days); OR Stabilized acute coronary syndrome (unstable angina (CCS III, or CCS IV), non STEMI, or STEMI with no chest pain or other cardiac symptoms for >24 hours
* Blood cardiac biomarker (i.e. troponin I, CK-MB) levels less than the local laboratory ULN within 12 hours of the time of PCI guidewire placement.
* Subject is to undergo PCI of a single lesion in a single native coronary artery during the enrollment procedure.
* There is prior intent to treat the target lesion as part of the patient's clinical care.
* The target lesion angiographic stenosis visually estimated as >=50% and <100%
* The target lesion reference vessel diameter must be >=2.5mm (visually estimated)
* Total target lesion length must be ≤60 mm (visually estimated)
* The minimum landing zone requirements for the FilterWire device can be met.
* There must be no major side branches (>2.0 mm in diameter) within the target lesion.
* There must be no major side branches (>2.0mm in diameter) between the target lesion and the filter nitinol loop landing zone.

Exclusion Criteria

* Subject is currently, or within the preceding 30 days, participating in a device or pharmaceutical treatment protocol.
* Subject life expectancy at time of enrollment is less than 2 years;
* Subject is pregnant or suspected to be pregnant at time of enrollment
* Prior coronary bypass graft surgery (CABG)
* PCI performed within the 24hours prior to the start of the study procedure
* A PCI is planned within the 30 days following the enrollment procedure.
* Unable to take aspirin and a thienopyridine for at least 30 days
* Patient experienced a STEMI or non STEMI within the past 24 hours
* Documented LVEF <25%
* the patient has multi-lesion or multi-vessel disease requiring revascularization of multiple lesions during the enrollment catheterization
* Any angiographic evidence of thrombus in any coronary artery
* There is evidence of dissection or procedural complication prior to randomization
* Patient has unprotected left main (≥50% stenosis) or left main equivalent disease
* Target Lesion is located in the distal segment of the target native coronary artery
* Proximal bound of the target lesion is located within 3mm of the ostium of the target vessel or major side branch (>2mm diameter by visual estimate)
* Target lesion is excessively calcified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evidence of Peri-procedural Myocardial Infarction as the result of standard care stenting procedure. | <24 hours after percutaneous coronary intervention
  The occurrence of a peri-procedural MI in the context of the CANARY trial will be defined as an elevation of troponin I (cTnI), or troponin T (cTnT) above three times the upper limit of normal (>3xULN).

SECONDARY OUTCOMES:
Evidence of Peri-procedural Myocardial Infarction as the result of standard | <24 hours after percutaneous coronary intervention
  The occurrence of a peri-procedural MI in the context of the CANARY trial will be defined as an elevation of creatine kinase myocardial band (CK-MB) biomarker above three times the upper limit of normal (>3xULN).
Frequency of Intraprocedural complications related to the treatment of the Target Plaque. | Catheterization Start Time to Completion Time.
  Instances of TIMI flow degradation, Procedural Success, Dissection/Perforations, abrupt closure, thrombus generation, etc will be recorded to determine the any gross differences in event rates between the study groups.
Composite MACE | from discharge from initial hospital stay to 30 (+/-7days) following the procedure
  The composite major adverse cardiac event rate (death, myocardial infarction, revascularization of the target lesion or vessel, cerebral vascualar accident will be reported for all groups at 30 days from the initial treatment (+/- 7 days).
Composite MACE | 365 days (+/- 30days) from initial procedure
  The composite major adverse cardiac event rate (death, myocardial infarction, revascularization of the target lesion or vessel, cerebral vascualar accident will be reported for all groups at 365 days from the initial treatment (+/- 30 days).

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W. Stone, M.D., Principal Investigator — Columbia University
Locations (9):
- United States (9):
  - Scottsdale Healthcare Shea, Scottsdale, Arizona
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Spectrum Health System, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mount Sinai School of Medicine Hospital, New York, New York
  - Pinnacle Health Cardiovascular Insititute, Harrisburg, Pennsylvania
  - Medical University of South Carolina Hospital, Charleston, South Carolina
  - Veterans Affairs North Texas Health Care Systems, Dallas, Texas